CLINICAL TRIAL: NCT02522494
Title: Encouraging Patient-Centered Communication in Clinical Video Telehealth Visits
Acronym: TELEHEALTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SDR 12-282
Record Dates: First submitted 2015-06-26; First posted 2015-08-13 (Estimated); Results first posted 2021-06-01 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Telemedicine; Videotape Recording

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Patients randomized to the intervention will view the video
  Interventions: Behavioral: Pamphlet; Behavioral: Video
- Pamphlet alone (Other): Patients randomized to the pamphlet alone will only receive the pamphlet
  Interventions: Behavioral: Pamphlet

INTERVENTIONS:
Behavioral: Pamphlet — An educational intervention delivered prior to patients' visits with primary care physicians.
  Other Names: Speak Up for Telehealth
Behavioral: Video — An educational intervention delivered prior to patients' visits with primary care providers.
  Other Names: Speak Up Video for Telehealth
  Arms: Intervention

SUMMARY:
Diabetes is common, it is expensive, and it is a chronic condition. Estimates put the prevalence of diabetes at almost 20 percent in VA patients. Poorly controlled diabetes leads to a number of complications including cardiovascular disease, blindness, amputation, and end stage renal disease. Adherence to medication regimens (as well as lifestyle factors such as diet and exercise) is important to achieve diabetes care goals. Adherence to recommended care is related at least in part to effective communication in medical encounters. This project is designed to test a video intervention to improve patients' communication behaviors. Providers will also receive a pamphlet with specific recommendation to improve communication skills. The project will assess the impact of the training programs on communication and outcomes. The study is designed to help make patient care more patient-centered, which is one of the six aims for improvement in the IOM Report, Crossing the Quality Chasm and is a goal of VA transformation efforts.

DETAILED DESCRIPTION:
Background: Clinical video telehealth (CVT) offers the opportunity for more efficient access to high quality primary and specialist care for Veterans. Enthusiasm for CVT is especially high in the VA given geographical separation between many Veterans and their providers at VA Medical Centers. However, because CVT encounters are by nature less personal than in-person visits, communication during CVT visits may be more challenging for both patients and providers resulting in less patient-centered communication. Less personal visits may have less exchange of information, lower satisfaction, less trust, and poorer outcomes. Indeed, research comparing CVT with in-person consultations found that patients in CVT visits were more passive and that CVT interactions were dominated by providers when compared with in-person visits.

This project will leverage prior work from two HSR&D-funded pilot projects to improve provider - patient communication for Veterans with type 2 diabetes mellitus. In a short-term project, SHP-08-182, the investigators conducted focus groups to elicit and understand patients' barriers to communicating with their providers. This qualitative work was used in a subsequent pilot project, PPO-08-402 to develop an educational video to encourage Veterans to use active participatory communication in their visits to providers. This work was successfully completed and the product is a 10-minute video that, in testing, was found to be acceptable and feasible to show to VA patients immediately preceding their medical encounters.

Objectives: The investigators goal in this project is develop and test a video intervention and to also develop pamphlets for patients and providers to encourage active and positive communication in CVT medical interactions. The investigators goal was developed with and is supported by the project's operational partner the Office of Telehealth Services and is integral to the goal to ensure patient-centered care in new models of care. Patient-centered communication in medical interactions is critical and plays an important, but often overlooked, role in the delivery of health services.

There are two aims. First, the investigators will develop educational interventions to encourage patients and providers to use active communication behaviors during CVT visits. Second, the investigators will conduct a randomized trial of the video and pamphlet (intervention) vs. pamphlet alone (comparison) in a two-arm randomized effectiveness trial. The investigators will evaluate for improvement in visit outcomes including patient and provider measures of patient-centered care and communication, reduction in several common barriers to clinical improvement, and improved medication adherence measures and hemoglobin A1c. In addition, the investigators will assess the mediators and moderators of the relationship of the intervention condition to outcomes.

Methods: The project will have two phases. In the initial phase of the proposed project the investigators will develop the video intervention. Video development will include qualitative interviews with stakeholders and patients regarding CVT barriers and perceived benefits. The investigators will use several existing resources and an expert panel of co-investigators and consultants to bring these elements together and produce the intervention. In phase 2 the investigators will conduct a randomized trial of the intervention, evaluating for improvement in a number of outcomes.

Impacts: The educational tools will be deliverables that could be used prior to CVT visits to improve communication and could serve as a paradigm for developing communication aids for other medical conditions and other clinical settings. The investigators will evaluate whether the educational intervention will help improve communication and will be associated with better visit and intermediate outcomes. Educational tools that encourage more patient-centered communication during CVT encounters may allow more rapid acceptance of CVT, thereby improving access to healthcare and enhancing the operational mission of the project's partner.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus,
* Hemoglobin A1c not controlled,
* Adults,
* Age 18 or older

Exclusion Criteria:

* Dementia,
* Lives in skilled nursing facility,
* Terminal medical condition,
* Drug-induced diabetes,
* Blind or deaf.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Gordon, MD BS, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (3):
- United States (3):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Jesse Brown VA Medical Center Community-Based Outpatient Clinic Lake Side Divison, Chicago, IL, Chicago, Illinois
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gopal RK, Solanki P, Bokhour BG, Skorohod N, Hernandez Lujan DA, Choi W, Gordon HS. Provider, Staff, and Patient Perspectives on medical Visits Using Clinical Video Telehealth: A Foundation for Educational Initiatives to Improve Medical Care in Telehealth. J Nurse Pract. 2021 May;17(5):582-587. doi: 10.1016/j.nurpra.2021.02.020. PMID 34471399
- [Derived] Gordon HS, Pugach O, Solanki P, Gopal RK. A brief pre-visit educational video improved patient engagement after telehealth visits; results from a randomized controlled trial. PEC Innov. 2022 Sep 5;1:100080. doi: 10.1016/j.pecinn.2022.100080. eCollection 2022 Dec. PMID 37213724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total number of patients enrolled in randomized trial - 102.
Groups:
- Intervention: Patients randomized to the intervention arm worked with educational materials: 1) they view the intervention video that encouraged patients to use active communication behaviors showing positive role models overcoming common communication challenges in CVT visit, and 2) they read the pamphlet that described how to use active communication behaviors in CVT visits Both educational materials (the video and pamphlet) had been mailed to the participants. The participants worked with the educational materials prior to their scheduled CVT visit.
- Pamphlet Alone: Patients randomized to the control arm only read the pamphlet. The same pamphlet as in the intervention group had been mailed to the control patients prior to their scheduled CVT visit.
Period: Overall Study
Arm/Group | Intervention | Pamphlet Alone
Started | 51 | 51
Post-CVT Visit Interview | 37 | 48
4-Week Follow Up | 37 | 46
Completed | 37 | 46
Not Completed | 14 | 5
Not completed — Lost to Follow-up | 6 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — CVT visit cancelled or no-show for CVT visit | 6 | 2
Not completed — Participant did not watch the video | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Pamphlet Alone | Total
Number analyzed (Participants) | 37 | 48 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 19 | 32
  >=65 years | 24 | 29 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8.37) | 65 (9.38) | 65 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 37 | 46 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 16 | 28
  Not Hispanic or Latino | 25 | 31 | 56
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 32 | 45 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 48 | 85

OUTCOME MEASURES:

1. Primary Outcome: HgbA1c
Description: HgbA1c is regarded as the standard laboratory measurement (blood test) for assessing the control of diabetes over approximately three months preceding the test. HgbA1c is usually checked several times a year in patients with poorly controlled diabetes.
Time Frame: At the baseline (Pre-CVT visit interview) and post-intervention (Post-CVT visit interview). All available values were restricted to one year before Baseline (Pre-Visit Interview) and from 30 days to 6 months past Post-CVT visit Interview.
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
percentage of glycated hemoglobin
  pre-CVT visit | 8.5 (1.76) | 8.5 (1.20)
  post-CVT visit | 7.99 (1.28) | 8.2 (1.26)

2. Primary Outcome: Communication Self-efficacy
Description: Communication Self-Efficacy (pre and post visit) is the degree to which a patient feels able to interact with his/her provider in order to provide information about problems, obtain desired information about diagnosis, treatment and prognosis, and participate in formulating a plan. The Perceived Efficacy in Physician-Patient Interactions scale (PEPPI) is a valid and reliable measure of patients' perceived self-efficacy in interacting with physicians (alpha 0.83). The short form of the PEPPI (PEPPI-5) has 5-items. Score on the PEPPI-5 ranges from 5-25. Higher scores reflect a better perceived self-efficacy in interacting with physicians.
Time Frame: At the baseline (Pre-CVT visit interview) and post-intervention (interview within one week past CVT visit)
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale
  pre-CVT visit | 22.81 (4.61) | 21.64 (5.94)
  post-CVT visit | 22.94 (4.76) | 22.75 (5.89)

3. Primary Outcome: Consultation Care Measure (CCM)
Description: Consultation Care Measure (CCM) assesses patient-centered care and patient-centered communication. Patients rate such factors as their providers' (1) communication and partnership, (2) personal relationship, (3) health promotion, (4) positive and clear approach to problem, (5) interest in effect on life on a 21-item scale, each item scores from 1 (strongly disagree) to 5 (strongly agree). Scores can range from 21 to 105. The higher scores mean a better patients' experiences with their provider.
Time Frame: post-intervention (interview within 1 week after CVT visit)
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale | 90.22 (16.30) | 84.08 (21.43)

4. Primary Outcome: Adherence (Self-reported)
Description: Self-reported adherence is measured using a brief questionnaire - a general measure of adherence to providers' recommendations and includes 5 items and is scored on a 6-level Likert-type scale ranging from "none of the time" to "all of the time". Scores range from 0-100 (after normalizing the standard 6-30 range) with higher numbers reflecting better adherence. Adherence using this measure is assessed with a brief telephone survey 4 weeks following the visit.
Time Frame: 4 weeks after the CVT visit
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale | 78.51 (21.53) | 75.98 (26.43)

5. Primary Outcome: Medication Adherence (MPR)
Description: Medication adherence will be assessed with a medication possession ratio (MPR) for diabetes medications.
Time Frame: 6 months
Population: The data was not collected because it was not possible to calculate useful medication possession ratios. Many patients in our study were on insulin which is a liquid and is not a unit dose. Further many patients take insulin on a sliding scale. Calculating the MPR was therefore not a useful measure in this study.
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Adherence at 1 Year
Description: Medication adherence will be assessed with a medication possession ratio (MPR) for diabetes medications.
Time Frame: 1 year
Population: as for outcome 5
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Consultation and Relational Empathy (CARE)
Description: Consultation and Relational Empathy (CARE) Measure - is a tool for measuring patients' perceptions of relational empathy in the consultation. In this 10-item questionnaire patients rate the statements about their doctor's understanding their concern, showing care, and etc. during the recent CVT visit on a scale from 1 to 5 where 1 is "poor" and 5 is "excellent". Scores can range from 10 to 50. The higher score means a better patient's perception of empathy in consultation.
Time Frame: Post-intervention (interview within one week past CVT visit)
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale | 44.65 (7.75) | 40.39 (10.73)

8. Primary Outcome: Communication Ratings
Description: The questionnaire assesses patients' ratings of their own participatory communication behavior and patients' ratings of their providers' communication. It is a 15-item scale with 3 sub-scales. Patients' ratings of their (1) providers' informativeness and the extent to which the patient understands that information (information sub-scale) are measured with 5-items; (2) patients' ratings that the provider values and respects them is measured with 5-items; and (3) patients' ratings of their own communication is measured with 5-items. This questionnaire has high internal consistency. The scale is scored from 1 (completely disagree) to 7 (completely agree). The total scores range from 15 to 105. The higher scores indicate a better quality of communication.
Time Frame: Post-intervention (interview within one week after CVT visit)
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale | 94.24 (13.54) | 88.67 (18.55)

9. Primary Outcome: Human Connection Scale
Description: Human Connection Scale is a 15-item questionnaire that measures the extent to which patient feel a sense of mutual understanding, caring, and trust with their physicians. The scale is a valid and reliable measure of therapeutic alliance between patients and their physicians. The score from 1 to 4 is used where 1 is "not at all" and 4 is "extremely". The scores range from 15 to 60. The higher scores indicate higher therapeutic alliance between patients and physicians.
Time Frame: At the baseline (Pre-CVT visit interview) and post-intervention (Post-CVT visit interview)
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale
  pre-CVT visit | 49.73 (13.19) | 49.28 (12.05)
  post-CVT visit | 52.44 (10.63) | 49.35 (12.77)

10. Primary Outcome: Resistance to Treatment Questionnaire (RTQ)
Description: Resistance to Treatment Questionnaire (RTQ) identifies the reasons for resistance to treatment and its intensity among patients with diabetes. 20-item questionnaire consists of four themes (lack of faith or dissatisfaction, emotional reasons, specific problems, factors connected to despair or failure) containing 5 items each; each item is scored from 1 (strongly disagree) to 5 (strongly agree). The scores range from 20 to 100. The higher scores mean more barriers to treatment (a worse outcome).
Time Frame: 4 weeks past CVT visit
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale | 42.59 (11.06) | 45.13 (13.99)

11. Secondary Outcome: Trust in Provider Questionnaire
Description: Trust in Provider is an important characteristic of provider-patient relationships and is assessed with a questionnaire. Trust is measured pre- and post-CVT visit using a 9-item measure. The scale is scored on a 7-point Likert scale using the anchors "strongly disagree" and "strongly agree". The scores range from 9 to 63. The higher scores mean a better trust in provider.
Time Frame: At the baseline (Pre-CVT visit interview) and post-intervention (interview within one week after CVT visit)
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale
  pre-CVT visit | 47.08 (14.63) | 45.00 (15.16)
  post-CVT visit | 53.27 (8.88) | 50.19 (11.76)

12. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction is assessed as the extent to which the patient is content with the relationship with her/his provider, in terms of the quality of information exchanged during medical encounters, and in terms of the demeanor of the provider toward the patient (courtesy, respectfulness, sensitivity, taking time and not being rushed). This is a 4-item survey, patient's satisfaction is scored from 1 (not at all satisfied) to 7 (extremely satisfied). The scores range from 5 to 35. The higher score indicates a better patient satisfaction.
Time Frame: four weeks after CVT visit
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale | 24.19 (3.98) | 23.35 (5.45)

13. Secondary Outcome: Participatory Decision-Making
Description: Participatory Decision-Making Style represents the degree to which providers involve patients in decision making. We measure patients' ratings of providers' participatory decision-making style using a 4-item scale evaluated by Heisler et al. in a study of veterans with diabetes. The authors found it to be associated with better patient understanding of diabetes and self-management practices. The survey scores how often provider involves patient in decision-making on a scale from 1 to 5, where 1 is "none of the time" and 5 is "all of the time". Scores range from 4 to 20. Higher scores mean a better outcome.
Time Frame: At the baseline (Pre-CVT visit interview) and post-intervention (Post-CVT visit interview)
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale
  pre-CVT visit | 16.68 (4.45) | 15.34 (5.34)
  post-CVT visit | 17.15 (4.76) | 15.06 (5.10)

14. Secondary Outcome: Diabetes Self-Efficacy
Description: The investigators used a 4-item scale to measure patients' confidence in their ability to manage their diabetes. The survey scores patients' perception of how well they can handle their diabetes on a scale from 1 to 7, where 1 is "not at all true" and 7 is "very true". The scores range from 4 to 28. The higher score is validated as a predictor of better glycemic control. The higher scores mean a better confidence in managing diabetes.
Time Frame: At the baseline (Pre-CVT visit interview) and post-intervention (interview within one week after CVT visit)
Population: Veterans with diabetes mellitus whose HbA1c ≥7 and whose primary care includes CVT visits at ECHCS or JBVAMC.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Pamphlet Alone
Number analyzed (Participants) | 37 | 48
units on a scale
  pre-CVT visit | 22.81 (4.61) | 21.64 (5.94)
  post-CVT visit | 22.94 (4.76) | 22.75 (5.89)

ADVERSE EVENTS:
Time Frame: From the baseline (Pre-CVT visit interview Visit 1) to the follow-up telephone interview (four weeks past Post-CVT visit), an average of 3 months per participant. Time frame varies depending on occurrence of patients' Clinical Video Telehealth visits with their physicians in routine clinical practice.
Arm/Group | Intervention | Pamphlet Alone
All-Cause Mortality (participants affected / at risk) | 0/37 | 1/48
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/48
Other Adverse Events (participants affected / at risk) | 0/37 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=37) | Pamphlet Alone (N=48)
death (General disorders) | NA | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT02522494/Prot_SAP_000.pdf